CLINICAL TRIAL: NCT02975713
Title: Progesterone Diurnal Rhythm During Ovarian Stimulation for IVF
Status: Terminated | Type: Observational
Why Stopped: no participants were recruited,study stopped
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Medical Director, ART Fertility Clinics LLC
Other Study IDs: 1609-ABU-070-HF
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Hyperstimulation
Keywords: P4,ART,IVF,FSH,LH,AMH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples extracted from the vein
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the influence of circadian rhythm on progesterone levels during follicular phase of natural cycle and during follicular phase of controlled ovarian stimulation during IVF.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the circadian rhythm of progesterone in a stimulated cycle. Sample size calculations show that the study needs to recruit 10 women to show any significant differences in progesterone secreted in the morning at 8 am compared to that secreted in the evening at 8 pm. We have increased the number of participants to 12 in order to compensate for any possible drop outs. The hormones FSH, LH, Progesterone and Estradiol will be measured at days 2/3, 8, 10 and 12 of a normal and stimulated cycle so that each patient serves as her own control.

This study will provide the basis to establish the optimal blood sampling time for progesterone measurement and to more accurately determine the cut-off level for progesterone for favourable pregnancy outcomes in ART.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF / ICSI - treatment
* Age ≥ 18 years and ≤ 35 years
* Ovarian reserve parameters in the adequate age - range, determined by Anti-Mullerian-Hormone (AMH) and Antral Follicle Count (AFC)(16)
* Able to understand the aim of the study and to provide consent
* Regular cycle (25-35 days)

Exclusion Criteria:

* Diagnosis of polycystic ovarian syndrome (PCOS) Rotterdam criteria
* Endometriosis stage 3 or 4 AFS
* Treatment with GnRH-analogues during the previous 6 months
* Intake of oral contraceptive pill (OCP) or any hormonal treatment during the last 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have to undergo IVF due to primary or secondary infertility.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Progesterone levels during follicular phase | 2-4 months
  The primary aim of this study is to determine the circadian rhythm of progesterone in a stimulated cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Human Mo Fatemi, Medical Director, Principal Investigator — IVI Middle East Clinic
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fatemi HM, Van Vaerenbergh I. Significance of premature progesterone rise in IVF. Curr Opin Obstet Gynecol. 2015 Jun;27(3):242-8. doi: 10.1097/GCO.0000000000000172. PMID 25811257
- [Background] Patton PE, Lim JY, Hickok LR, Kettel LM, Larson JM, Pau KY. Precision of progesterone measurements with the use of automated immunoassay analyzers and the impact on clinical decisions for in vitro fertilization. Fertil Steril. 2014 Jun;101(6):1629-36. doi: 10.1016/j.fertnstert.2014.02.037. Epub 2014 Mar 21. PMID 24661729
- [Result] Venetis CA, Kolibianakis EM, Bosdou JK, Tarlatzis BC. Progesterone elevation and probability of pregnancy after IVF: a systematic review and meta-analysis of over 60 000 cycles. Hum Reprod Update. 2013 Sep-Oct;19(5):433-57. doi: 10.1093/humupd/dmt014. Epub 2013 Jul 4. PMID 23827986
- [Result] Huang R, Fang C, Xu S, Yi Y, Liang X. Premature progesterone rise negatively correlated with live birth rate in IVF cycles with GnRH agonist: an analysis of 2,566 cycles. Fertil Steril. 2012 Sep;98(3):664-670.e2. doi: 10.1016/j.fertnstert.2012.05.024. Epub 2012 Jun 15. PMID 22704632
- [Result] Ochsenkuhn R, Arzberger A, von Schonfeldt V, Gallwas J, Rogenhofer N, Crispin A, Thaler CJ, Noss U. Subtle progesterone rise on the day of human chorionic gonadotropin administration is associated with lower live birth rates in women undergoing assisted reproductive technology: a retrospective study with 2,555 fresh embryo transfers. Fertil Steril. 2012 Aug;98(2):347-54. doi: 10.1016/j.fertnstert.2012.04.041. Epub 2012 May 24. PMID 22633265
- [Result] Xu B, Li Z, Zhang H, Jin L, Li Y, Ai J, Zhu G. Serum progesterone level effects on the outcome of in vitro fertilization in patients with different ovarian response: an analysis of more than 10,000 cycles. Fertil Steril. 2012 Jun;97(6):1321-7.e1-4. doi: 10.1016/j.fertnstert.2012.03.014. Epub 2012 Apr 10. PMID 22494924
- [Result] Labarta E, Martinez-Conejero JA, Alama P, Horcajadas JA, Pellicer A, Simon C, Bosch E. Endometrial receptivity is affected in women with high circulating progesterone levels at the end of the follicular phase: a functional genomics analysis. Hum Reprod. 2011 Jul;26(7):1813-25. doi: 10.1093/humrep/der126. Epub 2011 May 2. PMID 21540246
- [Result] Van Vaerenbergh I, Fatemi HM, Blockeel C, Van Lommel L, In't Veld P, Schuit F, Kolibianakis EM, Devroey P, Bourgain C. Progesterone rise on HCG day in GnRH antagonist/rFSH stimulated cycles affects endometrial gene expression. Reprod Biomed Online. 2011 Mar;22(3):263-71. doi: 10.1016/j.rbmo.2010.11.002. Epub 2010 Nov 13. PMID 21273126
- [Result] Bosch E, Labarta E, Crespo J, Simon C, Remohi J, Jenkins J, Pellicer A. Circulating progesterone levels and ongoing pregnancy rates in controlled ovarian stimulation cycles for in vitro fertilization: analysis of over 4000 cycles. Hum Reprod. 2010 Aug;25(8):2092-100. doi: 10.1093/humrep/deq125. Epub 2010 Jun 10. PMID 20539042
- [Result] Kyrou D, Popovic-Todorovic B, Fatemi HM, Bourgain C, Haentjens P, Van Landuyt L, Devroey P. Does the estradiol level on the day of human chorionic gonadotrophin administration have an impact on pregnancy rates in patients treated with rec-FSH/GnRH antagonist? Hum Reprod. 2009 Nov;24(11):2902-9. doi: 10.1093/humrep/dep290. Epub 2009 Aug 11. PMID 19671625
- [Result] Strott CA, Yoshimi T, Lipsett MB. Plasma progesterone and 17-hydroxyprogesterone in normal men and children with congenital adrenal hyperplasia. J Clin Invest. 1969 May;48(5):930-9. doi: 10.1172/JCI106052. PMID 4305376
- [Result] Bungum L, Jacobsson AK, Rosen F, Becker C, Yding Andersen C, Guner N, Giwercman A. Circadian variation in concentration of anti-Mullerian hormone in regularly menstruating females: relation to age, gonadotrophin and sex steroid levels. Hum Reprod. 2011 Mar;26(3):678-84. doi: 10.1093/humrep/deq380. Epub 2011 Jan 11. PMID 21227943
- [Result] Bungum L, Franssohn F, Bungum M, Humaidan P, Giwercman A. The circadian variation in Anti-Mullerian hormone in patients with polycystic ovary syndrome differs significantly from normally ovulating women. PLoS One. 2013 Sep 4;8(9):e68223. doi: 10.1371/journal.pone.0068223. eCollection 2013. PMID 24023708
- [Result] Seifer DB, Baker VL, Leader B. Age-specific serum anti-Mullerian hormone values for 17,120 women presenting to fertility centers within the United States. Fertil Steril. 2011 Feb;95(2):747-50. doi: 10.1016/j.fertnstert.2010.10.011. Epub 2010 Nov 13. PMID 21074758